CLINICAL TRIAL: NCT02345525
Title: The Feasibility of a Home-based Constraint-Induced Movement Therapy Program in Chronic Stroke Survivors.
Brief Title: Constraint-Induced Movement Therapy in Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Studio CIMT
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mCIMT (Active Comparator): 2 hours intensive upper limb practice with shaping techniques supervised by an experienced physiotherapist + 2 hours ADLs at home (supervised by a caregiver) Patients are supposed to wear a mitt on the unaffected hand for 4 hours daily.
  Interventions: Behavioral: mCIMT
- hCIMT (Experimental): 2 hours intensive upper limb practice with shaping techniques + 2 hours ADLs supervised by a caregiver.
  Patients are supposed to wear a mitt on the unaffected hand for 4 hours daily.
  Interventions: Behavioral: hCIMT

INTERVENTIONS:
Behavioral: mCIMT — This intervention is based on 3 main aspects:
  1. intensive training of functional tasks with the affected arm (massed practice)
  2. constraint of the un-affected hand through a mitt
  3. shaping techniques designed to transfer gains to the real world activities
  The 2 hours massed practice will be performed in a outpatient clinic with a supervision of PT.
  Arms: mCIMT
Behavioral: hCIMT — This intervention is based on 3 main aspects:
  1. intensive training of functional tasks with the affected arm (massed practice)
  2. constraint of the un-affected hand through a mitt
  3. shaping techniques designed to transfer gains to the real world activities
  In this group, a comprehensive set of the material necessary to perform the training at home and a booklet containing an explanation of the exercises that can be done will be provided to subjects.
  In addition, 2 hospital visits will be scheduled to instruct subjects and caregivers on the training and to update activities (1 visit at the beginning + 1 visit after 1 week).
  Arms: hCIMT

SUMMARY:
The aim of this study is to evaluate the feasibility of a Home-based Constraint-Induced Movement Therapy (hCIMT) compared to a Modified Constraint-Induced Movement Therapy (mCIMT) delivered in a outpatient setting on upper limb motor recovery in stroke survivors.

DETAILED DESCRIPTION:
Home-based Constraint Induced Modified Therapy (hCIMT) consist of 2 hours intensive upper limb practice with shaping techniques + 2 hours ADLs supervised by a caregiver. Patients are supposed to wear a mitt on the unaffected hand for 4 hours daily.

Modified Constraint Induced Modified Therapy (mCIMT) consist of 2 hours intensive upper limb practice with shaping techniques supervised by an experienced physiotherapist + 2 hours ADLs at home (supervised by a caregiver) Patients are supposed to wear a mitt on the unaffected hand for 4 hours daily.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years and < 80 years
* diagnosis of first ischemic stroke
* stroke onset > 6 months prior to study enrollment
* upper extremity hemiparesis with impairment of hand and/or arm:
* active wrist extension ≥20º
* active metacarpophalangeal- and interphalangeal-joints extension ≥ 10°
* muscle tone assessed by the Modified Ashworth Scale (MAS) ≤ 2
* pain assessed by the Visual Analogue Scale (VAS) <4

Exclusion Criteria:

* anyone who does not have adequate understanding of verbal or written information in Italian sufficient to complete any test
* impaired cognitive functioning: score less than 24 on the Mini Mental Status Examination (MMSE)
* contraindications to single-pulse transcranial magnetic stimulation (TMS)(TMS will be used to measure cortical excitability): presence of a history of epilepsy, frequent headaches or neck pain, implantable devices (ventriculoperitoneal shunts, pacemakers, intrathecal pumps, intracranial metal implants)
* neurological or psychiatric pathology
* severe cardio-pulmonary, renal, hepatic diseases
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-08; Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in Fugl-Meyer Upper Extremity (FM-UE) | 1)A week prior to treatment beginning 2) the week after the end of treatment 4) at 3 months follow-up
  Measure of upper extremity motor impairment. The upper extremity score ranges from 0-66.

SECONDARY OUTCOMES:
Wolf Motor Function Test (WMFT) | 1)A week prior to treatment beginning 2) the week after the end of treatment 4) at 3 months follow-up
  Quantitative measure of upper extremity motor ability through timed and functional tasks.
Nine Hole Peg Test (NHPT | 1)A week prior to treatment beginning 2) the week after the end of treatment 4) at 3 months follow-up
  Measures finger dexterity
Motor Activity Log (MAL) | 1)A week prior to treatment beginning 2) the week after the end of treatment 4) at 3 months follow-up
  Assessment of the change in real-world arm use in activities of daily living. Subjects are asked to score the quality of movement as well as amount of use of the affected arm in a number of common daily activities.
Stroke Impact Scale 3.0 (SIS 3.0) | 1)A week prior to treatment beginning 2) the week after the end of treatment 4) at 3 months follow-up
  Self-assessment questionnaire assesses health status following stroke
Motor cortex excitability (single pulse and paired pulse TMS) | 1)A week prior to treatment beginning 2) the week after the end of treatment 4) at 3 months follow-up
  Single-Pulse TMS will be used to study cortical-spinal tract excitability in primary motor cortex (M1).
  Paired-pulse TMS Paired-Pulse TMS will be used to study intracortical excitability.
NIRS (Near Infrared Spectroscopy) NIRS measurements will be performed during 6 cycles of 15s hand reaching and grasping and 45s resting while sitting on a chair. | 1)A week prior to treatment beginning 2) the week after the end of treatment 4) at 3 months follow-up
  For the NIRS it will use an 32-channel NIRS imaging equipment which consist of 16 pairs of emitting and detecting optical fibers attached to a custom-made head cap placed on primary motor cortex.
  NIRS measurements will be performed during 6 cycles of 15s hand reaching and grasping and 45s resting while sitting on a chair.

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Straudi, MD, Principal Investigator — Ospedale San Giorgio
Locations (1):
- Ferrara University Hospital, Ferrara, Italy